CLINICAL TRIAL: NCT04256590
Title: Tongue Depressor-related Tongue Swelling in Adenoidectomy Surgeries in Pediatric Patients
Brief Title: Tongue Depressor-related Tongue Swelling
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Merih Onal, Assistant Professor, Selcuk University
Other Study IDs: 2018/18
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Children, Only; Adenoidal Hypertrophy; Adenoid Disease - Chronic; Complication; Side Effect
Keywords: children; tongue disease; ultrasonography; enlarge tongue; adenoid
MeSH Terms: conditions — Tongue Diseases | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study: Patients aged 16 years or younger who were to undergo adenoidectomy surgery were eligible for inclusion in this group. Tongue surface areas were measured twice by submental USG.The first measurements (TSA2) were done immediately after endotracheal intubation but before insertion and placement of the tongue depressor. The second measurements (TSA1) were done after adenoidectomy surgery and after removal of the tongue depressor but just before extubation. The difference between TSA2 and TSA1 (i.e., (TSA2-TSA1) was used to defined the occurrence of tongue swelling.
  Interventions: Diagnostic Test: Ultrasonography imaging
- Control: This group included patients aged 16 years or younger who did not need adenoidectomy surgery and any head and neck procedures. Tongue surface areas of the patients were measured twice by submental USG as in the study group. TSA1s were done immediately after endotracheal intubation, and TSA2s were done at the end of the surgical procedure just before extubation. The difference between TSA2 and TSA1 (i.e., (TSA2-TSA1) was used to defined the occurrence of tongue edema.
  Interventions: Diagnostic Test: Ultrasonography imaging

INTERVENTIONS:
Diagnostic Test: Ultrasonography imaging — This study aimed to measure the tongue surface areas of the patients two times both of study and control groups with ultrasonography imaging to compare the tongue surface areas.

SUMMARY:
This study aimed to detect tongue swelling induced by the pressure exerted by tongue depressor; swelling detection was made through tongue surface area measurement using ultrasonography (USG) in pediatric patients who underwent adenoidectomy surgeries.

DETAILED DESCRIPTION:
The tongue is an ideal organ for ultrasonography (USG) evaluation. This study aimed to detect the occurrence of tongue swelling through USG examination and to educate clinicians about the association between subacute tongue swelling and tongue depressor in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 years or younger
* Undergo adenoidectomy surgery
* Patients informed consent obtained from the parents

Inclusion Criteria for control group:

* Patients aged 16 years or younger
* Patients who did not need adenoidectomy surgery and any head and neck procedures
* Patients who underwent endotracheal intubation under general anesthesia except adenoidectomy and head and neck surgery.

Exclusion Criteria:

* Patients aged older than 16 years
* Patients with a history of syndromal craniofacial abnormalities
* Patients with systemic disorders and other otolaryngologic problems

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 16 years or younger who were to undergo adenoidectomy surgery were eligible for inclusion in this group. Informed consent was obtained from the parents of all the patients with a clinical diagnosis of chronic adenoiditis and adenoid hypertrophy (except tonsillectomy surgeries) and were to undergo adenoidectomy surgery.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change from preoperative measurement to postoperative measurement in tongue surface area on the ultrasonography imaging. | 2018-2019 (6 months)
  This study aimed to evaluate the change from baseline in tongue surface area on the ultrasonography imaging due to the tongue depressor.

SECONDARY OUTCOMES:
Detection of swelling formation in tongue by using ultrasonography imaging. | 2018-2019 (6 months)
  This study aimed to measure and detect the tongue swelling by using ultrasonography imaging due to the tongue depressor.

CONTACTS AND LOCATIONS:
Overall Officials: Merih Onal, Principal Investigator — Selcuk University
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)